CLINICAL TRIAL: NCT06694194
Title: Global, Regional, and National Burdens and Trends of Tracheal, Bronchial, and Lung Cancer in Individuals Aged 70 Years and Older from 1990 to 2021
Acronym: GDBlung70
Status: Completed | Type: Observational
Sponsor: Hongquan Xing (Other)
Responsible Party: Sponsor-Investigator, Hongquan Xing, M.D, Nanchang University
Organization: Nanchang University (Other)
Other Study IDs: NanchangUN
Record Dates: First submitted 2024-11-11; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 1990-01

CONDITIONS: Lung Cancer Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The incidence, mortality, and disability-adjusted life years (DALYs) data for TBL cancer patients aged ≥ 70 years, spanning 1990-2021, were sourced from the 2021 Global Burden of Disease (GBD) study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NA

SUMMARY:
Despite the increasing health burden of tracheal, bronchial, and lung (TBL) cancer patients aged ≥ 70 years worldwide, data on its burden and trends are limited. This study aimed to analyze the global, regional, and national burdens and trends of TBL cancer from 1990 to 2021.

DETAILED DESCRIPTION:
The latest cancer report indicates that tracheal, bronchial, and lung (TBL) cancer, the most widespread cancer globally, accounts for 12.4% of new diagnoses and 18.7% of cancer-related deaths, thereby presenting significant societal, public health, and economic challenges.Despite the increasing health burden of tracheal, bronchial, and lung (TBL) cancer patients aged ≥ 70 years worldwide, data on its burden and trends are limited. This study aimed to analyze the global, regional, and national burdens and trends of TBL cancer from 1990 to 2021.

ELIGIBILITY:
Inclusion Criteria:

Pathologic Diagnosis of lung cancer

Exclusion Criteria:

breast cancer Age less than 70 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with lung cancer and aged 70 years and older
Sampling Method: Non-Probability Sample
Enrollment: 111627 (Actual)
Dates: Start 1990-01-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
The incidence, mortality, and disability-adjusted life years (DALYs) data for TBL cancer patients aged ≥ 70 years, spanning 1990-2021. | 1990-2021
  We extracted the incidence, mortality, and disability-adjusted life years (DALYs) for TBL cancer in individuals aged ≥ 70 years and above along with their 95% uncertainty intervals (UIs) from the GBD 2021 database (https://vizhub.healthdata.org
  /gbd-results/). The data were stratified by age groups and social determinants of the health index (SDI) regions, encompassing 21 global GBD regions and 204 countries.